CLINICAL TRIAL: NCT03987776
Title: The Effect of an Anti-Inflammatory Diet on Weight Loss, Body Composition, Cardiometabolic Risk Factors and Immune System Response in Younger Adults
Brief Title: An Anti-inflammatory Diet Effect on Metabolic, Inflammatory and Immune Status of Obese Younger Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center Rijeka (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, Sanja Klobučar Majanović, Assistant Professor, Clinical Hospital Center Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AIDIETOBESITY18-269/441
Record Dates: First submitted 2019-06-10; First posted 2019-06-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: anti-inflammatory diet; obesity; low-grade inflammation; cardiometabolic; immunity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The randomized controlled intervention study. A nutritional intervention will be based on an energy-restricted anti-inflammatory diet that will be compared with an isocaloric standard diet (55-60% carbohydrates, 25% fat, 15-20% protein).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory diet (Experimental): energy-reduced diet with the use of low glycemic foods, wholegrain products, legumes, colorful vegetables and fruit, nuts, seeds, marine fish, olive oil, green/black tea, and multiple spices and herbs
  Interventions: Behavioral: Anti-inflammatory energy-restricted diet
- Control energy-resticted diet (Experimental): isocaloric to anti-inflammatory diet, energy restricted diet (55-60% carbohydrates, 25% fat, 15-20% protein) used in a standard obesity management
  Interventions: Behavioral: Control energy-restricted diet

INTERVENTIONS:
Behavioral: Anti-inflammatory energy-restricted diet — During 6 months the participants will we asked to use recommended energy-reduced diet with anti-inflammatory properties, based on colorful vegetables and fruits, legumes, nuts, seeds, marine fish, whole-grain products, and daily use of olive oil, green/black tea, multiple spices and herbs.
  Arms: Anti-inflammatory diet
Behavioral: Control energy-restricted diet — During 6 months the participants of control group will be asked to use recommended energy-reduced diet based on standard obesity management (55-60% carbohydrates, 25% fat, 15-20% protein)
  Arms: Control energy-resticted diet

SUMMARY:
Diet has a major role in the etiology of obesity, and there is a growing body of evidence suggesting that a variety of dietary factors can modulate obesity-induced chronic low-grade inflammation and thus the course of obesity-related chronic non-communicable diseases. The present intervention study aims to evaluate the effect of an anti-inflammatory diet on weight loss, body composition, cardiometabolic risk factors and immune system response among young adults of the obese younger adults.

DETAILED DESCRIPTION:
Obesity pandemic presents a major challenge to chronic disease prevention worldwide. A low-grade chronic inflammation is associated with obesity and related cardiometabolic disorders, such as cardiovascular diseases, type 2 diabetes and some type of cancers. Diet has a major role in the etiology of obesity, and there is a growing body of evidence suggesting that a variety of dietary factors can modulate obesity-induced chronic low-grade inflammation and thus the course of obesity-related chronic non-communicable diseases. The present intervention study aims to evaluate the effect of an anti-Inflammatory diet on weight loss, body composition, cardiometabolic risk factors and immune system response among younger adults. A nutritional intervention based on an energy-restricted anti-inflammatory diet will be compared with an isocaloric standard diet (55-60% carbohydrates, 25% fat, 15-20% protein). The inflammatory potential of the diet will be assessed with the Dietary Inflammatory Index®.

ELIGIBILITY:
Inclusion Criteria:

* adults age of 18 to 50 years
* body mass index ≥ 30 kg/m2
* with or without obesity related complications

Exclusion Criteria:

* smoking
* chronic hearth, renal and/or liver diseases,
* active carcinoma or having carcinoma in last year
* anti-inflammatory and/or immunosuppressive drugs intake
* changing the existing medication therapy
* persons older than 50 years
* active infection and/or surgical procedure in last 3 months
* nutritive allergy or intolerance to any anti-inflammatory diet constituent
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
The changes in the body mass index | baseline, follow up 6 months
  body mass index (kg/m2) calculated from measured body weight (kg) and height (m)
The changes in the waist circumference | baseline, follow up 6 months
  waist circumference (cm) measured with measuring tape
The changes of fat mass | baseline, follow up 6 months
  fat mass (kg) measured with bioelectric impedance analyzer
The changes of fat-free mass | baseline, follow up 6 months
  fat-free mass (kg) measured with bioelectric impedance analyzer
The changes of skeletal muscle mass | baseline, follow up 6 months
  skeletal muscle mass (kg) measured with bioelectric impedance analyzer
The changes of visceral adipose tissue | baseline, follow up 6 months
  visceral adipose tissue (l) measured with bioelectric impedance analyzer

SECONDARY OUTCOMES:
The changes in fasting glucose concentration | baseline, follow up 6 months
  concentration of fasting glucose (mmol/l)
The changes in HbA1c concentration | baseline, follow up 6 months
  concentration of HbA1c (mmol/mol; %)
The changes in insulin concentration | baseline, follow up 6 months
  concentration of insulin (mU/l)
The changes of HOMA-index | baseline, follow up 6 months
  concentration of insulin (pmol/l) and glucose (mmol/l) for calculation of HOMA-index: HOMA - IR = (insulin (mU/l) x glucose (mmol/l)) / 22,5
The changes in serum lipid profile | baseline, follow up 6 months
  concentration of fasting triglycerides (mmol/l), HDL (mmol/l), LDL (mmol/l), total cholesterol (mmol/l)
The changes in serum liver transaminases concentration | baseline, follow up 6 months
  concentration of serum fasting liver transaminases (AST (U/l), ALT (U/l), GGT (U/l), ALP (U/l))
The changes in serum IL-beta, IL-6 and TNF-alpha concentrations | baseline, follow up 6 months
  concentration of serum IL-1 beta (pg/ml), IL-6 (pg/ml), TNF-alpha (pg/ml)
The changes in serum hs-C-reactive protein concentration | baseline, follow up 6 months
  concentration of serum hs-C-reactive protein (mg/l)
The changes of blood lymphocytes T and lymphocite subgroups count | baseline, follow up 6 months
  count of blood lymphocytes T, lymphocyte subgroups (TCD3, TCD4, TCD8, BCD19, NKCs, Tregs (CD4+CD25+Foxp3+))
The changes in thyroid stimulating hormone (TSH) concentration | baseline, follow up 6 months
  concentration of TSH (mIU/l)
The changes in free tri-iodothyronine (fT3) concentration | baseline, follow up 6 months
  concentration of fT3 (pmol/l)
The changes in free thyroxine (fT4) concentration | baseline, follow up 6 months
  concentration of fT4 (pmol/l) and thyroid peroxidase antibodies concentration (IU/l)
The changes in thyroid peroxidase antibodies (TPOAbs) concentration | baseline, follow up 6 months
  concentration of TPOAbs (IU/l)

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Klobučar Majanović, A. Prof., Principal Investigator — Clinical Hospital Centre Rijeka; Ines Mrakovčić Šutić, Prof., Principal Investigator — University of Rijeka, Faculty of Medicine; Gordana Kenđel Jovanović, Mag.nutr., Principal Investigator — Teaching Institute of Public Health of Primorsko-goranska County
Locations (1):
- Clinical Hospital Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Yes
We planned to share the statistical analysis results of the study, after the study will be completed and published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available one year after ending of the study for an year.

REFERENCES:
- [Background] Gonzalez-Muniesa P, Martinez-Gonzalez MA, Hu FB, Despres JP, Matsuzawa Y, Loos RJF, Moreno LA, Bray GA, Martinez JA. Obesity. Nat Rev Dis Primers. 2017 Jun 15;3:17034. doi: 10.1038/nrdp.2017.34. PMID 28617414
- [Background] Salas-Salvado J, Diaz-Lopez A, Ruiz-Canela M, Basora J, Fito M, Corella D, Serra-Majem L, Warnberg J, Romaguera D, Estruch R, Vidal J, Martinez JA, Aros F, Vazquez C, Ros E, Vioque J, Lopez-Miranda J, Bueno-Cavanillas A, Tur JA, Tinahones FJ, Martin V, Lapetra J, Pinto X, Daimiel L, Delgado-Rodriguez M, Matia P, Gomez-Gracia E, Diez-Espino J, Babio N, Castaner O, Sorli JV, Fiol M, Zulet MA, Bullo M, Goday A, Martinez-Gonzalez MA; PREDIMED-Plus investigators. Effect of a Lifestyle Intervention Program With Energy-Restricted Mediterranean Diet and Exercise on Weight Loss and Cardiovascular Risk Factors: One-Year Results of the PREDIMED-Plus Trial. Diabetes Care. 2019 May;42(5):777-788. doi: 10.2337/dc18-0836. Epub 2018 Nov 2. PMID 30389673
- [Background] Netea MG, Balkwill F, Chonchol M, Cominelli F, Donath MY, Giamarellos-Bourboulis EJ, Golenbock D, Gresnigt MS, Heneka MT, Hoffman HM, Hotchkiss R, Joosten LAB, Kastner DL, Korte M, Latz E, Libby P, Mandrup-Poulsen T, Mantovani A, Mills KHG, Nowak KL, O'Neill LA, Pickkers P, van der Poll T, Ridker PM, Schalkwijk J, Schwartz DA, Siegmund B, Steer CJ, Tilg H, van der Meer JWM, van de Veerdonk FL, Dinarello CA. A guiding map for inflammation. Nat Immunol. 2017 Jul 19;18(8):826-831. doi: 10.1038/ni.3790. PMID 28722720
- [Background] Schipper HS, Prakken B, Kalkhoven E, Boes M. Adipose tissue-resident immune cells: key players in immunometabolism. Trends Endocrinol Metab. 2012 Aug;23(8):407-15. doi: 10.1016/j.tem.2012.05.011. Epub 2012 Jul 12. PMID 22795937
- [Background] Satyaraj E. Emerging paradigms in immunonutrition. Top Companion Anim Med. 2011 Feb;26(1):25-32. doi: 10.1053/j.tcam.2011.01.004. PMID 21435623
- [Background] Salama AA, Amine EK, Salem HA, Abd El Fattah NK. Anti-Inflammatory Dietary Combo in Overweight and Obese Women with Polycystic Ovary Syndrome. N Am J Med Sci. 2015 Jul;7(7):310-6. doi: 10.4103/1947-2714.161246. PMID 26258078
- [Background] Mayr HL, Itsiopoulos C, Tierney AC, Ruiz-Canela M, Hebert JR, Shivappa N, Thomas CJ. Improvement in dietary inflammatory index score after 6-month dietary intervention is associated with reduction in interleukin-6 in patients with coronary heart disease: The AUSMED heart trial. Nutr Res. 2018 Jul;55:108-121. doi: 10.1016/j.nutres.2018.04.007. Epub 2018 Apr 25. PMID 29807669
- [Background] Turner-McGrievy GM, Wirth MD, Shivappa N, Dunn CG, Crimarco A, Hurley TG, West DS, Hussey JR, Hebert JR. Impact of a 12-month Inflammation Management Intervention on the Dietary Inflammatory Index, inflammation, and lipids. Clin Nutr ESPEN. 2019 Apr;30:42-51. doi: 10.1016/j.clnesp.2019.02.008. Epub 2019 Mar 1. PMID 30904228
- [Background] Sears B. Anti-inflammatory diets for obesity and diabetes. J Am Coll Nutr. 2009 Aug;28 Suppl:482S-491S. doi: 10.1080/07315724.2009.10718115. PMID 20234036
- [Background] Ricker MA, Haas WC. Anti-Inflammatory Diet in Clinical Practice: A Review. Nutr Clin Pract. 2017 Jun;32(3):318-325. doi: 10.1177/0884533617700353. Epub 2017 Mar 28. PMID 28350517
- [Background] Agarwal AK. Spice up your life: adipose tissue and inflammation. J Lipids. 2014;2014:182575. doi: 10.1155/2014/182575. Epub 2014 Feb 20. PMID 24701352
- [Background] Jiang TA. Health Benefits of Culinary Herbs and Spices. J AOAC Int. 2019 Mar 1;102(2):395-411. doi: 10.5740/jaoacint.18-0418. Epub 2019 Jan 16. PMID 30651162
- [Background] Rubio L, Motilva MJ, Romero MP. Recent advances in biologically active compounds in herbs and spices: a review of the most effective antioxidant and anti-inflammatory active principles. Crit Rev Food Sci Nutr. 2013;53(9):943-53. doi: 10.1080/10408398.2011.574802. PMID 23768186
- [Background] Ramirez AG, Parma DL, Munoz E, Mendoza KD, Harb C, Holden AEC, Wargovich M. An anti-inflammatory dietary intervention to reduce breast cancer recurrence risk: Study design and baseline data. Contemp Clin Trials. 2017 Jun;57:1-7. doi: 10.1016/j.cct.2017.03.009. Epub 2017 Mar 22. PMID 28342988
- [Background] Winkvist A, Barebring L, Gjertsson I, Ellegard L, Lindqvist HM. A randomized controlled cross-over trial investigating the effect of anti-inflammatory diet on disease activity and quality of life in rheumatoid arthritis: the Anti-inflammatory Diet In Rheumatoid Arthritis (ADIRA) study protocol. Nutr J. 2018 Apr 20;17(1):44. doi: 10.1186/s12937-018-0354-x. PMID 29678183
- [Background] McMorrow AM, Connaughton RM, Magalhaes TR, McGillicuddy FC, Hughes MF, Cheishvili D, Morine MJ, Ennis S, Healy ML, Roche EF, Tremblay RE, Szyf M, Lithander FE, Roche HM. Personalized Cardio-Metabolic Responses to an Anti-Inflammatory Nutrition Intervention in Obese Adolescents: A Randomized Controlled Crossover Trial. Mol Nutr Food Res. 2018 May;62(10):e1701008. doi: 10.1002/mnfr.201701008. PMID 29665620
- [Background] Yannakoulia M, Poulimeneas D, Mamalaki E, Anastasiou CA. Dietary modifications for weight loss and weight loss maintenance. Metabolism. 2019 Mar;92:153-162. doi: 10.1016/j.metabol.2019.01.001. Epub 2019 Jan 6. PMID 30625301
- [Background] Bianchi VE. Weight loss is a critical factor to reduce inflammation. Clin Nutr ESPEN. 2018 Dec;28:21-35. doi: 10.1016/j.clnesp.2018.08.007. Epub 2018 Sep 3. PMID 30390883
- [Background] Medina-Remon A, Casas R, Tressserra-Rimbau A, Ros E, Martinez-Gonzalez MA, Fito M, Corella D, Salas-Salvado J, Lamuela-Raventos RM, Estruch R; PREDIMED Study Investigators. Polyphenol intake from a Mediterranean diet decreases inflammatory biomarkers related to atherosclerosis: a substudy of the PREDIMED trial. Br J Clin Pharmacol. 2017 Jan;83(1):114-128. doi: 10.1111/bcp.12986. Epub 2016 May 19. PMID 27100393
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Tabung F, Hebert JR. A population-based dietary inflammatory index predicts levels of C-reactive protein in the Seasonal Variation of Blood Cholesterol Study (SEASONS). Public Health Nutr. 2014 Aug;17(8):1825-33. doi: 10.1017/S1368980013002565. Epub 2013 Oct 10. PMID 24107546
- [Background] Namazi N, Larijani B, Azadbakht L. Dietary Inflammatory Index and its Association with the Risk of Cardiovascular Diseases, Metabolic Syndrome, and Mortality: A Systematic Review and Meta-Analysis. Horm Metab Res. 2018 May;50(5):345-358. doi: 10.1055/a-0596-8204. Epub 2018 May 3. PMID 29723899
- [Background] Hebert JR, Shivappa N, Wirth MD, Hussey JR, Hurley TG. Perspective: The Dietary Inflammatory Index (DII)-Lessons Learned, Improvements Made, and Future Directions. Adv Nutr. 2019 Mar 1;10(2):185-195. doi: 10.1093/advances/nmy071. PMID 30615051
- [Background] Kendel Jovanovic G, Mrakovcic-Sutic I, Pavicic Zezelj S, Susa B, Rahelic D, Klobucar Majanovic S. The Efficacy of an Energy-Restricted Anti-Inflammatory Diet for the Management of Obesity in Younger Adults. Nutrients. 2020 Nov 22;12(11):3583. doi: 10.3390/nu12113583. PMID 33266499
- [Background] Kendel Jovanovic G, Pavicic Zezelj S, Klobucar Majanovic S, Mrakovcic-Sutic I, Sutic I. Metabolic syndrome and its association with the Dietary Inflammatory Index (DII)(R) in a Croatian working population. J Hum Nutr Diet. 2020 Feb;33(1):128-137. doi: 10.1111/jhn.12695. Epub 2019 Oct 11. PMID 31602707